CLINICAL TRIAL: NCT06758557
Title: A Multicenter, Open Phase Ib/II Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of HB0025 Injection Combined With Chemotherapy in Patients With Advanced Solid Tumor
Brief Title: A Study to Evaluate the Safety and Efficacy of HB0025 Injection in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Collaborators: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB0025-C-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-03 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Advanced NSCLC; Advanced Endometrial Cancer
Keywords: NSCLC; Endometrial Cancer; Clinical Trial
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Pemetrexed; Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: Sequential Assignment This study will enroll no more than 36 subjects at 10mg/kg and 20mg/kg respectively every 3 weeks (Q3W) in NSCLC and EC Cohort in phase Ib, no exceed 18 subjects in each Cohort, to compare the safety and efficacy, and will be extended to the group with better efficacy and tolerance.
  In the dose expansion phase(Phase II), 40 subjects will be enrolled in each expansion cohort. For advanced NSCLC groups, dose expansion of 4 cohorts at 2 dose levels are planned while 2 cohorts at 2 dose levels are in advanced EC groups. The study protocol may also be revised based on the interim data and dose expansion of 6 cohorts at 3 dose levels will be carried out in advanced NSCLC groups and 3 cohorts at 3 dose levels will be in advanced EC groups.
  In the Phase II expansion phase, 240 subjects are planned to be enrolled. In the Phase Ib/II study, no more than 282 subjects will be enrolled in total.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 10 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC (Experimental): 10 mg/kg of HB0025 combined Pemetrexed 500 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in Non-sq-NSCLC, with:
  (a)tyrosine kinase inhibitor (TKI) drug sensitivity mutations of epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) translocation, who have experienced disease progression after standard treatment with TKI targeted drugs, or are intolerant to standard treatment with TKI targeted drugs(for Phase Ib) or(b) with no previous systemic anti-tumor treatment(for Phase II).
  Interventions: Drug: HB0025; Drug: Pemetrexed; Drug: Carboplatin
- 20 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC (Experimental): 20 mg/kg of HB0025 combined Pemetrexed 500 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in Non-sq-NSCLC, with tyrosine kinase inhibitor (TKI) drug sensitivity mutations of epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) translocation, who have experienced disease progression after standard treatment with TKI targeted drugs, or are intolerant to standard treatment with TKI targeted drugs.
  Interventions: Drug: HB0025; Drug: Pemetrexed; Drug: Paclitaxel
- 10 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer (Experimental): 10 mg/kg of HB0025 combined Paclitaxel 175 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in EC, with no previous systemic anti-tumor treatment.
  Interventions: Drug: HB0025; Drug: Paclitaxel; Drug: Carboplatin
- 20 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer (Experimental): 20 mg/kg of HB0025 combined Paclitaxel 175 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in EC, with no previous systemic anti-tumor treatment.
  Interventions: Drug: HB0025; Drug: Paclitaxel; Drug: Carboplatin
- 10 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC (Experimental): 10 mg/kg of HB0025 combined Paclitaxel175 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in Non-sq-NSCLC, with no previous systemic anti-tumor treatment(for Phase II).
  Interventions: Drug: HB0025; Drug: Paclitaxel; Drug: Carboplatin
- 20 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC (Experimental): 20 mg/kg of HB0025 combined Paclitaxel 175 mg/m² iv d1+Carboplatin AUC 5 iv d1 in the patient in Non-sq-NSCLC, with no previous systemic anti-tumor treatment(for Phase II)
  Interventions: Drug: HB0025; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: HB0025 — HB0025 IV every 3 weeks (q3w)
Drug: Pemetrexed — 500 mg/m² iv d1
  Arms: 10 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC; 20 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC
Drug: Paclitaxel — 175 mg/m² iv d1
  Arms: 10 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC; 10 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer; 20 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC; 20 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer; 20 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC
Drug: Carboplatin — AUC 5 iv d1
  Arms: 10 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC; 10 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer; 10 mg/kg HB0025+Pemetrexed+Carboplatin for safety and intolerance in Non-sq-NSCLC; 20 mg/kg HB0025+Paclitaxel+Carboplatin for safety and intolerance in sq-NSCLC; 20 mg/kg HB0025+Paclitaxel+Carboplatin, for safety and intolerance in endometrial cancer

SUMMARY:
This study is a multicenter, two-tumor, multi-cohort, dose-escalation and dose-expansion Phase Ib/II clinical trial of HB0025 combined with chemotherapy, consists of two phases: the dose escalation phase (Ib) and the dose expansion phase (II).

1. The dose escalation phase (Phase Ⅰb) The primary purpose is to determine the Maximum Tolerated Dose(MTD) and/or dose limiting toxicity (DLT) of HB0025 combined with chemotherapy. The dose escalation is carried out using the "3+3 dose escalation" principle. In the initial stage of the dose escalation process, the chemotherapy dose remains unchanged to explore the safety and tolerability of the currently confirmed safe doses of HB0025 as monotherapy at 10mg/kg, and 20mg/kg, combined with chemotherapy(Pemetrexed 500 mg/m² iv d1+Carboplatin AUC 5 iv d1) in the treatment of advanced non-squamous non-samll cell lung cancer(Non-sq-NSCLC), and combined with chemotherapy( Paclitaxel 175 mg/m² iv d1+ Carboplatin AUC 5 iv d1 ) in advance Endometrial carcinoma(EC).

   After completing the first cycle of treatment (DLT evaluation period), if the investigator determines that the subject may benefit from the combined treatment, the subject will continue the treatment cycles (2nd to 4th/5th/6th cycle of HB0025 combined with chemotherapy); if there is no disease progression and no intolerable toxicity, the subject can continue to receive the maintenance treatment with HB0025 + pemetrexed (for non-sq NSCLC) or HB0025 alone (for EC, sq NSCLC), until when intolerable toxicity occurs, disease progression, the subject is lost to follow-up or died, the subject withdraws informed consent, the subject receives other anti-tumor treatment or the study is terminated early, whichever occurs first.
2. Dose expansion phase (Phase II) Based on 1-2 recommended Phase II doses selected by the sponsor and the investigator during the dose escalation process, a multicenter, single-arm study will be conducted to evaluate the efficacy and safety of different doses of HB0025 combined with chemotherapy. Each dosing regimen cohort will be expanded by 40 subjects. If a dosing regimen is not safe or effective, the enrollment of the dosing regimen cohort may be stopped, and the subject quota may be allocated to other dosing regimen cohorts (which may exceed 40 subjects). The dose expansion phase initially plans to expand the following cohorts to further observe the safety of HB0025 combined with chemotherapy and the preliminary efficacy of HB0025 combined with chemotherapy in advanced NSCLC and EC.

After receiving 4-6 cycles of HB0025 combined with chemotherapy, the subjects will enter HB0025 + pemetrexed (for non-sq-NSCLC) or HB0025 alone (for EC, sq-NSCLC) maintenance treatment until when intolerable toxicity, disease progression or death occurs, withdraw informed consent, or receives other anti-tumor treatment or study ends early, early, whichever occurs first.

DETAILED DESCRIPTION:
The design of dose level and Cohorts:

Phase Ib:

Advanced Non-sq-NSCLC(dose escalation phase):

The dose level of HB0025 including the following leves, the dose of chemotherapy is fixed(Pemetrexed 500 mg/m² iv d1+Carboplatin AUC 5 iv d1) in the study.

dose 1: 10mg/kg, dose 2: 20mg/kg, dose -1: 6mg/kg, dose +1: 15mg/kg, dose +2: 30mg/kg.

Advanced EC and sq-NSCLC:

With the same dose level design above, HB0025 combined with Paclitaxel(175 mg/m² iv d1) and Carboplatin(AUC 5 iv d1) in the treatment of advanced EC and sq-NSCLC.

Phase II:

Advanced non-small cell lung cancer indications:

1. Cohort 1: Patients with recurrent, metastatic, locally advanced non-squamous non-small cell lung cancer (Non-sq-NSCLC) who have not received systemic anti-tumor treatment and do not carry EGFR sensitive mutations or ALK fusion gene sensitive mutations; HB0025 at 10mg/kg combined with Pemetrexed 500 mg/m² iv d1 + Carboplatin AUC 5 iv d1; expended to approximately 40 subjects.
2. Cohort 2: Patients with recurrent, metastatic, locally advanced Non-sq-NSCLC who have not received systemic anti-tumor treatment and do not carry EGFR sensitive mutations or ALK fusion gene sensitive mutations; HB0025 at 20mg/kg combined with the same dose as cohort 1; expended to approximately 40 subjects.
3. Cohort 3: Patients with recurrent, metastatic, locally advanced squamous non-small cell lung cancer (Sq-NSCLC) who have not received systemic anti-tumor treatment and do not carry EGFR sensitive mutations or ALK fusion gene sensitive mutations; HB0025 at 10mg/kg combined with Paclitaxel 175mg/m² iv d1 + Carboplatin AUC 5 iv d1; expanded to approximately 40 subjects.
4. Cohort 4: Patients with recurrent, metastatic, locally advanced Sq-NSCLC who have not received systemic anti-tumor treatment and do not carry EGFR sensitive mutations or ALK fusion gene sensitive mutations; HB0025 at 20 mg/kg combined with the same dose as Cohort 3; extended to approximately 40 subjects.

Advanced endometrial cancer indications:

1. Cohort 1: Patients with recurrent, metastatic, locally advanced endometrial cancer who have not received systemic anti-tumor treatment before; HB0025 at 10 mg/kg combined with Paclitaxel 175 mg/m² iv d1 + Carboplatin AUC 5 iv d1; expanded to approximately 40 subjects.
2. Cohort 2: Patients with recurrent, metastatic, locally advanced endometrial cancer who have not received systemic anti-tumor treatment before; HB0025 at 20mg/kg combined with chemotherapy as the same dose as Chort1; expanded to approximately 40 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age between 18-75 years old (include 18- and 75-year-old);
2. Be able to fully understand and voluntarily sign the informed consent form, and be willing and able to comply with the clinical research and follow-up visit procedures；
3. Dose escalation phase 3.1 Non-small cell lung cancer and meet all following conditions； 3.1.1 Non-small cell lung cancer (NSCLC) confirmed by histology or cytology; 3.1.2 Not suitable for surgical resection, recurrence, metastasis, or locally advanced stage; 3.1.3 Patients with tyrosine kinase inhibitor (TKI) drug sensitivity mutations of epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) translocation, who have experienced disease progression after standard treatment with TKI targeted drugs, or are intolerant to standard treatment with TKI targeted drugs; 3.1.4 No known ROS proto-oncogene 1 (ROS1), neurogenic tyrosine receptor kinase (NTRK), proto-oncogene B-raf (BRAF), RET mutations or other oncogenic driver gene mutations, and there are approved therapeutic drugs for the above gene mutations (there are therapeutic drugs for genomic changes).

   3.2 Endometrial cancer and meet all following conditions 3.2.1 Endometrial cancer confirmed by histology or cytology, the pathological types include but are not limited to endometrioid carcinoma, serous carcinoma, clear cell carcinoma, undifferentiated carcinoma, dedifferentiated carcinoma, mixed carcinoma, and carcinosarcoma; 3.2.2 Not suitable for surgical resection, recurrence, metastasis, locally advanced stage; 3.2.3 No previous systemic anti-tumor treatment (excluding adjuvant therapy and neoadjuvant therapy);
4. Dose expansion phase 4.1 Non-small cell lung cancer and meet all following conditions 4.1.1 Non-squamous non-small cell lung cancer (Nonsq-NSCLC) or squamous non-small cell lung cancer (Sq-NSCLC) confirmed by histology or cytology (for central squamous cell carcinoma, the investigator and the sponsor jointly decide whether to enroll based on the risk of bleeding and the benefit-risk ratio of the subject); 4.1.2 Not suitable for surgical resection, recurrent, metastatic, locally advanced; Negative for TKI drug sensitivity mutations of epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) translocation; 4.1.3 Negative for TKI drug sensitivity mutations of epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK) translocation; 4.1.4 No known ROS proto-oncogene 1 (ROS1), neurogenic tyrosine receptor kinase (NTRK)，proto-oncogene B-raf (BRAF), RET mutations or other oncogenic driver gene mutations, for which there are approved therapeutic drugs for the above gene mutations (there are therapeutic drugs for genomic changes); 4.1.5 No previous systemic anti-tumor treatment (for subjects who have received adjuvant/neoadjuvant treatment for non-metastatic disease with the purpose of cure, if disease progression occurs within 6 months of the end of the last treatment, the treatment regimen is considered as one systemic treatment and is not allowed to be included).

   4.2 Endometrial cancer and meet all following conditions 4.2.1 Endometrial cancer confirmed by histology or cytology, with pathological types including but not limited to endometrioid carcinoma, serous carcinoma, clear cell carcinoma, undifferentiated carcinoma, dedifferentiated carcinoma, mixed carcinoma, and carcinosarcoma; 4.2.2 Not suitable for surgical resection, recurrence, metastasis, locally advanced stage; 4.2.3 No previous systemic anti-tumor treatment (for subjects who have received adjuvant/ neoadjuvant treatment for non-metastatic disease with the purpose of cure, if disease progression occurs within 6 months of the end of the last treatment, the treatment regimen is considered as 1 systemic treatment and is not allowed to be included in the group);
5. Patients who have not received anti-tumor treatment or other clinical trial drugs within 4 weeks before the first administration of HB0025 (for small molecule targeted drugs, this is within 2 weeks before the first use of the study drug or within 5 half-lives of the drug (whichever is longer); have completed systemic palliative radiotherapy for at least 4 weeks or local palliative radiotherapy for at least 2 weeks (in the baseline tumor assessment, the target lesions defined can be excluded if they are not in the local radiotherapy area); have not systematically used (for 2 consecutive weeks) traditional Chinese medicine with anti-tumor indications within 2 weeks before the first use of the study drug;
6. There is at least one measurable tumor lesion (according to RECIST 1.1 standard); Note: Lesions that have been previously treated with local therapy (e.g., radiofrequency ablation, anhydrous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound, trans-arterial chemoembolization, local radiotherapy, etc.) are not considered measurable lesions unless there is clear progression.
7. ECOG score of 0 or 1;
8. The expected survival period is not less than 12 weeks;
9. The following laboratory indicators must be met:

   9.1 Absolute neutrophil count ≥1.5×10⁹/L; 9.2 Platelet count ≥90×10⁹/L; 9.3 Hemoglobin ≥90 g/L; Note: The above three requirements require that the patient has not received any blood component or cell growth factor support therapy within two weeks before blood collection.

   9.4 Creatinine clearance ≥50 mL/min (Cockcroft-Gault Formula); 9.5 Total bilirubin ≤1.5×ULN; 9.6 Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤2.5× ULN; If the investigator determines that the increase is due to liver metastasis of the tumor, ALT和AST≤5×ULN; 9.7 Prothrombin time (PT)≤1.5×ULN, partial thromboplastin time (APTT)≤1.5×ULN; 9.8 Urine dipstick test results show protein in urine<1+; if urine protein ≥1+, 24-hour urine protein content<1 g.
10. The toxicity from previous treatment has recovered to grade 1 (except for toxicity such as alopecia that the investigator determines does not pose a safety risk);
11. Females and males of childbearing age must agree to take effective contraceptive measures during the study and within 3 months after the last dose of HB0025 after signing the informed consent form. Female subjects of childbearing age must have a negative pregnancy test result during the screening period.

Exclusion Criteria:

1. Brain metastasis with central nervous system symptoms; for subjects with asymptomatic brain metastasis: after receiving relevant treatment, imaging and neurological examinations are in a stable state for more than 4 weeks. If there is no imaging evaluation, the neurological examination is in a stable state for more than 4 weeks under glucocorticoid treatment, and the treatment dose for at least 2 weeks is ≤10mg/day of prednisone or other hormones of the same dose, they can be included in the group;
2. Active autoimmune diseases or a history of autoimmune diseases requiring systemic treatment within 2 years before screening, including hypothyroidism, Graves' ophthalmo-pathy, Hashimoto's thyroiditis or type 1 diabetes, but childhood asthma or allergic asthma that did not occur within 2 years before screening can be excluded;
3. Patients who received >10 mg/day of prednisone or equivalent dose of systemic glucocorticoids or other immunosuppressants within 2 weeks before screening, or who received topical, intraocular, intraarticular, intranasal or inhaled hormones for prevention (such as contrast agent allergy) or treatment of non-autoimmune diseases (such as delayed hypersensitivity reactions caused by contact allergens) were allowed to be included in the group;
4. Any of the following infections:

   4.1 Active infection within 2 weeks prior to screening, requiring antibiotic treatment for >7 days; 4.2 Active pulmonary tuberculosis (based on history); 4.3 HIV positive; 4.4 Active hepatitis B or hepatitis C. Asymptomatic hepatitis B virus carriers (HBV DNA titer below the detection limit) or clinically cured hepatitis C (HCV RNA test negative) are allowed to enroll;
5. Patients who have received immune checkpoint inhibitors (ICI) combined with anti-vascular therapy, such as anti-PD-(L)-1 antibody combined with anti-VEGF, VEGFR antibody, or TKI drugs with anti-vascular effects such as anlotinib;
6. Patients with a history of severe allergies, previous grade 3-4 immune-related adverse events (irAEs) or treatment discontinuation (except for grade 3 endocrine abnormalities that can be controlled by hormone replacement therapy); patients with grade 3-4 allergic reactions when receiving other monoclonal antibody treatments, or patients with known allergies to protein drugs or recombinant proteins, HB0025 drug components, and chemotherapy drug components;
7. Uncontrolled arterial hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment;
8. Suffering from the following serious comorbidities:

   8.1 Subjects with a history of arterial thrombosis or deep vein thrombosis within 6 months before screening, or subjects with evidence or history of bleeding tendency within 2 months before enrollment, regardless of severity (For the EC cohort: the decision on whether to enroll subjects with evidence or history of bleeding tendency within 2 months before enrollment was made by the investigator and the sponsor); 8.2 Previous or current bleeding or coagulation disorders; 8.3 Past history of myocarditis, cardiomyopathy, or malignant arrhythmias. Clinically significant (e.g., active) cardiovascular and cerebrovascular diseases within 6 months prior to screening, including but not limited to unstable angina requiring hospitalization, myocardial infarction, New York Heart Association-classified congestive heart failure ≥ II, severe arrhythmias that cannot be controlled by drugs, transient ischemic attack (TIA), cerebrovascular accident (CVA) or vascular disease (e.g., aortic aneurysm with risk of rupture), or other cardiac damage that may affect the safety evaluation of the study drug (e.g., poorly controlled arrhythmias, myocardial ischemia), etc.; 8.4 Gastrointestinal disorders or conditions that may cause gastrointestinal bleeding or perforation (history of intestinal obstruction, acute Crohn's disease, ulcerative colitis, esophageal varices, unhealed ulcers, unhealed wounds, intra-abdominal abscesses, or acute gastrointestinal bleeding within 6 months prior to screening). Subjects with chronic Crohn's disease and ulcerative colitis (except those with total colon and rectal resection), even in the inactive stage, should be excluded; 8.5 Those who have had digestive tract perforation or fistula, urogenital system fistula, and have not recovered after surgical treatment; 8.6 Current clinically significant hydronephrosis that has not been relieved by nephrostomy or ureteral stenting; 8.7 Patients with third space effusion (such as pleural effusion, pericardial effusion or ascites) that is currently clinically poorly controlled and requires repeated puncture drainage or other local treatment; 8.8 Imaging (CT or MRI) shows that the tumor has invaded or surrounded important blood vessels (lung cancer cohort only) or the investigators judge that the tumor is very likely to invade important blood vessels and cause fatal bleeding during the follow-up study; 8.9 Acute exacerbation of COPD within 1 month before first dose;
9. Patients who have used or are currently taking anticoagulants such as warfarin, heparin (except for tube sealing and deep vein catheterization), dabigatran etexilate, rivaroxaban, etc. within 7 days before the first study treatment; or patients who have received aspirin, clopidogrel, dipyridamole, cilostazol, or other drugs known to inhibit platelet aggregation;
10. Received major surgical treatment, open biopsy or significant trauma within 4 weeks before drug administration; or required major elective surgical treatment during the study period. Received local invasive procedures (such as needles) within 1 week before drug administration. Core biopsy), except for placement of a vascular access device;
11. Those with past and/or current interstitial lung disease, pneumoconiosis, drug-related pneumonia, severe lung function impairment, etc. that may interfere with the detection and treatment of suspected drug-related pulmonary toxicity;
12. Pregnant or breastfeeding women;
13. History of allogeneic organ transplantation or hematopoietic stem cell transplantation;
14. Second tumor within 5 years before screening, excluding cured cervical cancer in situ, localized skin squamous cell carcinoma, basal cell carcinoma, breast ductal carcinoma in situ or T1 urothelial carcinoma;
15. Received live virus vaccine within 30 days before screening;
16. During the screening period, patients with advanced Nonsq-NSCLC who are intolerant to the chemotherapy regimen of pemetrexed combined with carboplatin;
17. During the screening period, patients with advanced sq-NSCLC or EC who are intolerant to paclitaxel combined with carboplatin chemotherapy;
18. Subjects who are assessed by the investigator to be unsuitable for participating in the trial due to other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 24 Months
  ORR defined as the number of patients were confirmed complete response(CR) and/or partial response(PR) according to RECIST 1.1 divided by the patients with at least one tumour evaluation

SECONDARY OUTCOMES:
Disease control rate (DCR) | up to 24 mouths
  DCR defined as the number of patients were confirmed CR and/or PR and/or stable disease(SD) according to RECIST 1.1 divided by the patients with at least one tumour evaluation
Overall survival (OS) | up to 24 months
  Overall survival is defined as the time from the start of treatment with HB0025 until death due to any cause. OS as evaluated by investigators according to RECIST v1.1
Duration of response (DOR) | up to 24 months
  DOR defined as time from the first record of CR or PR to the first record of tumor progression or death of subjects
Progression-free Survival（PFS） | up to 24 months
  progression-free survival (PFS) means the time between the start of treatment and the onset of tumor progression or death from various causes.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | up to 24 months
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Maximum serum concentration(Cmax) | up to 24 months
  Cmax refers to The maximum blood concentration of HB0025 after administration. Sample concentration analysis method adopts ELISA.
Half-life (t1/2) | up to 24 months
  t1/2 refers to the time of a half reduction of total drug concentration in the body. parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
time of maximum concentration(Tmax) | Up to 24 Months
  Peak time after HB0025 administration. The parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis
Maximum serum concentration(Cmax) | up to 24 months
  Cmax refers to The maximum blood concentration of HB0025 after administration. - Sample concentration analysis method adopts ELISA . - parameters will be calculated by Phoenix WinNonlin version 8.3 using non-compartmental analysis.
Anti-drug antibodies (ADA) | up to 24 months
  Incidence of positive anti-drug antibodies(ADA)

CONTACTS AND LOCATIONS:
Overall Officials: Caicun Zhou, PhD., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China; Jundong Li, PhD., Principal Investigator — Sun Yat-sen University
Locations (14):
- China (14):
  - Affiliated Hospital of Hebei University / School of Clinical Medicine, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First People'S Hospital of Lianyungãng, Lianyungang, Jiangsu
  - Liaoning Cancer Hospital＆Institute, Shenyang, Liaoning
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Weifang People'S Hospital, Weifang, Shandong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer hospital, Taiyuan, Shanxi
  - The First Affiliated Hospitalof Xi'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospitalzhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No